CLINICAL TRIAL: NCT00849043
Title: A Single Arm, Open-label Extension Study to Evaluate the Long-term Durability of Treatment Response and and Safety of the Provent Professional Sleep Apnea Therapy Device for the Non-invasive Treatment of Obstructive Sleep Apnea-hypopnea
Brief Title: Extension Study of Original Protocol AERO C009 for Obstructive Sleep Apnea-hypopnea
Acronym: AERO C009E
Status: Completed | Type: Observational
Sponsor: Ventus Medical, Inc. (Industry)
Responsible Party: Connie Rey, Ventus Medical, Inc
Other Study IDs: AERO C009E
Record Dates: First submitted 2009-02-19; First posted 2009-02-23 (Estimated); Last update posted 2011-01-26 (Estimated); Status verified 2011-01

CONDITIONS: Obstructive Sleep Apnea Hypopnea; Obstructive Sleep Apnea; OSAH
Keywords: obstructive sleep apnea hypopnea; OSA; OSAH
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Provent: Provent Professional Sleep Apnea Therapy device

SUMMARY:
The purpose of this study is to evaluate the long-term durability of the treatment and safety of the Provent device for those individuals who were enrolled in the C009 study, were diagnosed with obstructive sleep apnea-hypopnea (OSAH), and were actively using the Provent device.

ELIGIBILITY:
Inclusion Criteria:

1. Based upon scoring at the study site, the 3-month 'device on' PSG has a 50% reduction in AHI compared to the 1-week 'device off' PSG AHI OR the 3-month 'device on' PSG AHI <10
2. Used the Provent device at least 4 hours for at least 5/7 nights per week on average during months 1 and 2 of the three month C009 study
3. The study physician and investigator believe that continued Provent use does not represent a significant safety risk for the patient
4. Patient understands and is willing and able to comply with study requirements

Exclusion Criteria:

1. The patient must continue to not meet all of the exclusion criteria of protocol C009

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: OSA subjects from C009 AERO study who were randomized to the Provent arm and completed the study. All must continue to meet the C009 inclusion and exclusion criteria.
Sampling Method: Probability Sample
Enrollment: 65 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To measure the percent change in the subject's apnea-hypopnea index (AHI) during the 12 month PSG while wearing the Provent device as compared to their AHI during the first week PSG when the subject did not wear the Provent device in the C009 study | 12 months

SECONDARY OUTCOMES:
Measurement of the subjects quality of life | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Meir Kryger, MD, Principal Investigator — Gaylord Sleep Medicine Research
Locations (13):
- United States (13):
  - Gaylord Sleep Medicine Research, Wallingford, Connecticut
  - University of Florida Health Science Center, Gainesville, Florida
  - Sleep Disorders Center of Georgia, Atlanta, Georgia
  - Suburban Lung Associates, Elk Grove Village, Illinois
  - Kentucky Research Group, Louisville, Kentucky
  - Sleep HealthCenters, Brighton, Massachusetts
  - Wayne State University Harper Univ. Hospital, Detroit, Michigan
  - Borgess Research, Kalamazoo, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - St. Luke's Hospital Sleep Medicine & Research Center, Chesterfield, Missouri
  - The Corvallis Clinic, Corvallis, Oregon
  - Sleep Medicine Associates of Texas, Dallas, Texas
  - Sleep Therapy and Research Center, San Antonio, Texas

REFERENCES:
- [Derived] Kryger MH, Berry RB, Massie CA. Long-term use of a nasal expiratory positive airway pressure (EPAP) device as a treatment for obstructive sleep apnea (OSA). J Clin Sleep Med. 2011 Oct 15;7(5):449-53B. doi: 10.5664/JCSM.1304. PMID 22003339